CLINICAL TRIAL: NCT01952249
Title: SIERRA: A Phase 1b/2 Study of Demcizumab Plus Paclitaxel in Subjects With Platinum Resistant Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: A Study of Demcizumab Plus Paclitaxel in Subjects With Platinum Resistant Ovarian
Acronym: SIERRA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase 2 portion not initiated, no longer pursuing ovarian cancer indication
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18-005
Record Dates: First submitted 2013-09-18; First posted 2013-09-27 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Primary Peritoneal Carcinoma
Keywords: Ovarian; Primary Peritoneal; Fallopian Tube Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — demcizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Demcizumab (Experimental): Demcizumab will be administered prior to paclitaxel by intravenous (IV) infusion.
  Interventions: Drug: Demcizumab; Drug: Taxol
- Taxol (Experimental): demcizumab combined with weekly paclitaxel
  Interventions: Drug: Demcizumab; Drug: Taxol

INTERVENTIONS:
Drug: Demcizumab — administered intravenously
  Other Names: OMP-21M18
Drug: Taxol — administered intravenously

SUMMARY:
This is a Phase 1b/2 study of paclitaxel plus demcizumab in subjects with platinum resistant ovarian, primary peritoneal or fallopian tube cancer.

DETAILED DESCRIPTION:
Phase 1b portion was completed; Phase 2 portion was not initiated.

Subjects must not have received prior weekly paclitaxel or more than 3 prior chemotherapy regimens in the Phase 1b portion of the study and more than 2 prior chemotherapy regimens in the Phase 2 portion of the study. Prior to enrollment, subjects will undergo screening to determine study eligibility. In the Phase 1b portion of study, 3 subjects will be treated at each dose level if no dose-limiting toxicities (DLTs) are observed. If 1 of 3 subjects experiences a DLT, that dose level will be expanded to 6 subjects.

If 2 or more subjects experience a DLT, no further subjects will be dosed at that level and 3 additional subjects will be added to the preceding dose cohort unless 6 subjects have already been treated at that dose level. Subjects will be assessed for DLTs from Days 0-28. Dose escalation for newly enrolled subjects, if appropriate, will occur after all subjects in a cohort have completed their Day 28 DLT assessment. After the final patient in the Phase 1b portion of the trial has completed their Day 28 DLT assessment, 50 subjects will be enrolled in the Phase 2 portion of the study and treated with demcizumab at the highest dose level that had < 2 DLTs in the 6 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have cytologically or histologically confirmed ovarian, primary peritoneal or fallopian tube cancer.. In addition, subjects must have a tumor that is at least 1 cm in a single dimension and is radiographically apparent on CT, PET-CT or MRI (i.e., RECIST version 1.1 measurable disease).
2. Subjects must have platinum resistant disease (i.e., which is defined as disease progression in less than 6 months after receiving a minimum of 4 cycles of a platinum containing regimen).
3. Subjects with the following histologic epithelial cell types are eligible: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma N.O.S.
4. Age >21 years
5. ECOG performance status <3

Exclusion Criteria:

1. Subjects receiving any other investigational medicinal product or anti-cancer therapy.
2. Prior therapy with weekly paclitaxel for recurrent disease (administration of weekly paclitaxel as part of an upfront treatment strategy is acceptable as long as the patient had not progressed while receiving weekly paclitaxel or recurred within 4 months of receiving weekly paclitaxel)
3. Non-epithelial ovarian carcinoma, including malignant mixed Mullerian tumors.
4. For the Phase 1b portion of the study, more than 3 prior chemotherapy regimens and for the Phase 2 portion of the study more than 2 prior chemotherapy regimens. Maintenance therapy following induction chemotherapy does not count as a separate regimen. In addition, hormonal therapy (e.g., tamoxifen or an aromatase inhibitor) does not count as a separate regimen.
5. Prior radiotherapy to the pelvis or abdomen
6. Subjects receiving heparin, warfarin, or other similar anticoagulants. Note: Subjects may be receiving lowdose aspirin and/or non-steroidal anti-inflammatory agents.

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Dose limiting toxicities (DLT) of demcizumab when combined with weekly paclitaxel in subjects with platinum resistant ovarian, primary peritoneal or fallopian tube cancer | Subjects will be treated and observed for DLT through the end of the first cycle (Days 0-28)
  The maximum tolerated dose (MTD) will be determined in patients treated with demcizumab in combination with weekly paclitaxel

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of demcizumab when given in combination with weekly paclitaxel | Plasma sample for Pharmacokinetics (PK) analysis to be obtained prior to the demcizumab infusion on Days 0, 14, 56 and 70 and at the end of the demcizumab infusion (prior to paclitaxel infusion) on Days 0 and 56.
  Apparent half life, AUC, clearance, volume of distribution

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center Department of Gynecologic Oncology, Houston, Texas